CLINICAL TRIAL: NCT04523597
Title: "Evaluation of Static and Dynamic Postural Balance in Children With Thoracic Hyperkyphosis"
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nazlı Elif Nacar, physical therapist, Istanbul University - Cerrahpasa
Other Study IDs: Istanbul University Cerrahpasa
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Hyperkyphosis
Keywords: Kyphosis; Postural Stability; Biodex Balance System; Equilibrium
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- toracic hyperkyphosis: children with COBB angle ≥ 45˚
- control: children with kyphosis index < 13 measured using the flexicurve ruler

SUMMARY:
The purpose of our study; is to investigate how balance parameters are affected in comparison with healthy children in children with thoracic hyperkyphosis and to examine the relationship of these results with muscle strength, shortness-flexibility, pain, range of motion, functional status, physical activity level and quality of life. The hypothesis of the study is that children with thoracic hyperkyphosis have impaired balance compared to their healthy peers. With this finding, it can be ensured that clinical evaluations and treatment strategies for balance in children with hyperkifosis are included in the treatment plan. 31 children with thoracic hyperkyphosis were included in the evaluation group, and 31 children with normal physiological curves were included in the control group. Participants were evaluated once by the physical therapist.

DETAILED DESCRIPTION:
The study was included chidren with hyperkyphosis at the İstanbul University-Cerrahpaşa, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation. G*Power 3.1.9.2 program was used to calculate the sample size. Due to the absence of MCID value for the Biodex Balance System in the literature while sample size calculation, the average values for males and females are 3.83 and 3.05 based on the "Overall Stability Index" based on the dominant side from a similar study conducted with healthy young adults; standard deviation values were placed in the formula as 1.03 and 1.13 (σ). (power=80%, α=0.05, significance level 2-tailed, and effect size d = 0.73). A total of 62 cases were decided to be included in the study, with 31 individuals per group. Participants were evaluated once by the physical therapist. Evaluation consist of demographic information form, Biodex Balance System, visual analog scale, "Hand-held" dynamometer, range of motion, pektoralis minor muscle flexibility, triple-hop distance test, 20-m sprint test, Physical Activity Questionnaire for Children, Pediatric Quality of Life Inventory, functional reach test and occiput-wall distance. SPSS (Statistical Package for Social Sciences) 22 statistical program was used for the statistical analysis of the data. Normality was assessed using the Shapiro-Wilk test. The "Chi-Square Test" was used to compare the difference between groups for categorical variables such as gender, dominant side, and educational status. The statistical analysis for group comparisons was performed using the "Mann-Whitney U Test" for non-parametric samples. Correlation analysis between the data was done with "Spearmann r Test". In all tests, a significance level of 0.05 (5%) was used.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic kyphosis angle: ≥ 45˚ (Cobb)
* Age between 9-18 years
* Volunteering to participate in the study
* Not physiotherapy
* Not cest tretment

Exclusion Criteria:

* Spinal surgery history
* Vision and hearing impairment
* Difficulty in detecting commands given
* Lower extremity affect that may affect balance
* Systemic disorder associated with balance
* Neurological influence
* > 20˚ (Cobb) scoliosis deformity

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children admitted to the orthopedics and Traumatology Outpatiant Clinic of Istanbul University, Istanbul Faculty of Medicine, and diagnosed with "thoracic Hypercyphosis" as a result of radiography evaluation.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Biodex Balance System | the cases were evaluated once.
  Biodex Balance System is a valid instrument used to measure postural stability in static and dynamic conditions. The stability platform allows for varying levels of difﬁculty of stability testing from level 1 (stabil) to level 12 (least stable). A high score is indicative of a lot of movement and indicates poor balance. In present study was assessed average Overall, AP, and ML stability scores under the following 4 position: right-leg static balance, left-leg static balance, bilateral static balance and bilateral dynamic balance at BBS level 8 (moderately unstable). Each position was applied with eyes open and closed.

SECONDARY OUTCOMES:
Visual Analog Scale | the cases were evaluated once.
  Visual Analogue Scale will be use to assess pain. The scale consists of a horizontal line between 0-100mm. A value of 0 mm indicates "no pain" and a value of 100 mm indicates "the most severe". The severity of the pain that the patients feel in the back and neck regions during rest, activity and at night will be evaluated numerically.
"Hand-held" dynamometer | the cases were evaluated once.
  Maximal isometric contraction was evaluated with "Hand-held" dynamometer (Lafeyette Instrument®, Lafayette, IN) using a standard protocol and recorded in kg / Newton. In our study, strength of trunk flexion and extansion, upper-middle-lower trapesiuz, serratus anterior, latissimus dorsi, bilateral hip flexion, extansion, abduction, knee flexion, extansion and ankle plantarflexion, dorsiflexion were examined bilaterally.
Range of Motion | the cases were evaluated once.
  Goniometric measurement is an objectively used method in the evaluation of ROM in the clinic. In our study, trunk flexion, extansion and lateral flexion were measured with goniometer.
Triple-Hop Distance (THD) test | the cases were evaluated once.
  Triple-Hop Distance test is considered to be a valid and reliable test in evaluating the functional status as it is easy to apply and does not require much time and equipment. Participants performed 3 consecutive maximal hops forward on the right and left limb. It was measured with tape the distance hopped from the starting line to the point where the heel struck the ground upon completing the third hop. The maximum distance achieved during the 3 trials was recorded in centimeters and was used for analysis. High scores indicate that the functional condition is good.
20-m sprint test | the cases were evaluated once.
  20-m sprint test is used to evaluate the maximum running time of the participants. Maximal effort sprint was assessed from a stationary start. Participants was instructed to stand with one foot right behind the starting line and to accelerate at maximum effort to the finish line. The best value of 3 trials (minimal sprint time) with a 2 min rest between trials was used for further data analysis. Time was taken with a stop watch.
Physical Activity Questionnaire for Children | the cases were evaluated once.
  The physical activity level of the participants wasevaluated with the Physical Activity Questionnaire for Children , which is frequently used in the clinic. This questionnaire consists of 9 items in the 5-point Likert type that questions the physical activities performed in the last 7 days and how often these activities are performed. A high score on the scale indicates that the physical activity level is high.
Pediatric Quality of Life Inventory | the cases were evaluated once.
  Pediatric Quality of Life Inventory is a quality-of-life scale with validity and reliability of 23 items, which are frequently used in research to question the quality of life in children and adolescents. The higher the score obtained from the scale, the higher the quality of life increases.
Functional reach test | the cases were evaluated once.
  It measures the distance (using a tape at the level of the acromion) that an participants are able to reach forward and sides from a starting standing position with a fixed base of support without loss of balance. In our study, the distance to the forward and sides of the cases was tested. For each position were made 3 measurements and their average values were calculated. High scores indicate that the functional balance is good.
The occiput-wall distance | the cases were evaluated once.
  The occiput-wall distance is a surrogate measure of kyphosis.The method has been verified for its reliability and validity. Two rulers were used to quantify the outcomes: the first ruler was placed on the landmark (occiput), and the second ruler was used to measure a perpendicular distance from the first ruler (occiput) to the wall. The measurement was repeated for three trials with a period of rest as needed between the trials, and the average distance over the three trials was used for the data analysis. Higher values indicate an increase in kyphosis angle.
muscle flexibility of pektoralis minor | the cases were evaluated once.
  The patients were placed in the supine position with their forearms pronated on the side of the body, in this position the distance between the acromion and the bed was measured with a tape measure and the value was recorded in cm. High values indicate muscle shortness.

CONTACTS AND LOCATIONS:
Overall Officials: Nazlı Nacar, Principal Investigator — Istanbul University-Cerrapaşa, Faculty of Health Sciences; Ayşe Zengin Alpözgen, Study Director — Istanbul University-Cerrapaşa, Faculty of Health Sciences
Locations (1):
- Istanbul University-Cerrapaşa, Faculty of Health Sciences, Istanbul, Turkey (Türkiye)